CLINICAL TRIAL: NCT00992537
Title: A Trial Comparing the Pharmacokinetic and Pharmacodynamic Properties Between NN5401 and NN1250 and Between NN5401 and Insulin Aspart in Subjects With Type 1 Diabetes
Brief Title: Comparison of the Effect of NN5401 With the Effect of NN1250 and Insulin Aspart in Type 1 Diabetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NN5401-1977; 2008-008357-32 (EudraCT Number); U1111-1111-9043 (Other: WHO)
Record Dates: First submitted 2009-10-08; First posted 2009-10-09 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — insulin degludec; insulin degludec, insulin aspart drug combination; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- IDeg (Experimental)
  Interventions: Drug: insulin degludec
- IDegAsp (Experimental)
  Interventions: Drug: insulin degludec/insulin aspart
- IAsp (Active Comparator)
  Interventions: Drug: insulin aspart

INTERVENTIONS:
Drug: insulin degludec — Insulin degludec single-dose of 0.5 U/kg body weight injected subcutaneously (under the skin).
  Arms: IDeg
Drug: insulin degludec/insulin aspart — Insulin degludec/insulin aspart single-dose of 0.5 U/kg body weight injected subcutaneously (under the skin).
  Arms: IDegAsp
Drug: insulin aspart — Insulin aspart single-dose of 0.5 U/kg body weight injected subcutaneously (under the skin).
  Arms: IAsp

SUMMARY:
This trial is conducted in Europe. The aim of this clinical trial is to compare the blood glucose lowering effect of NN5401(insulin degludec/insulin aspart (IDegAsp)) with NN1250 (insulin degludec (IDeg)) and insulin aspart (IAsp) in subjects with type 1 diabetes where the trial participant will receive one single dose of each trial product in varying order.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus (as diagnosed clinically) for at least 12 months
* Body mass index 18.0-28.0 kg/m^2 (both inclusive)

Exclusion Criteria:

* Subject who has donated any blood or plasma in the past month or more than 500 mL within 3 months prior to screening
* Smoker (defined as a subject who is smoking more than 5 cigarettes or the equivalent per day).
* Not able or willing to refrain from smoking and use of nicotine gum or transdermal nicotine patches during the inpatient period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2009-10; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Area under the glucose infusion rate curve | From 0 to 6 hours after single-dose administration
Area under the glucose infusion rate curve | From 4 to 24 hours after single-dose administration

SECONDARY OUTCOMES:
Area under the insulin degludec concentration-time curve | From 0 to 120 hours after single-dose administration
Maximum observed insulin degludec concentration | From 0 to 120 hours after single-dose administration
Area under the insulin aspart concentration-time curve | From 0 to 12 hours after single-dose administration
Maximum observed insulin aspart concentration | 0-12 hours after single-dose administration

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Neuss, Germany

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com